CLINICAL TRIAL: NCT04843215
Title: A Phase III, Multicenter, Prospective, Randomized, Controlled Clinical Trial Comparing Total and Partial Omentectomy for Patients With Advanced Gastric Cancer (TOP-GC)
Brief Title: A Phase III Study Comparing Total and Partial Omentectomy for Patients With Advanced Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Shanghai Zhongshan Hospital (Other); Fujian Cancer Hospital (Other Government); Fujian Medical University Union Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Harbin Medical University (Other); Hebei Medical University Fourth Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Changzhi People's Hospital (Other); The First Affiliated Hospital of Air Force Medicial University (Other); First Affiliated Hospital of Kunming Medical University (Other); LanZhou University (Other); Liaoning Cancer Hospital & Institute (Other); The First Affiliated Hospital of Nanchang University (Other); Shandong Provincial Hospital (Other Government); West China Hospital (Other); Xinjiang Medical University Cancer Hospital (Unknown); Zhejiang Cancer Hospital (Other); Chinese PLA General Hospital (Other); Sun Yat-sen University Cancer Hosptial (Unknown); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20210171
Record Dates: First submitted 2021-04-11; First posted 2021-04-13 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-04

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Prognosis; Omentectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group/D2 radical gastrectomy with partial omentectomy (Experimental): Partial omentectomy with preservation of the greater omentum at >3 cm from the gastroepiploic arcade.
  Interventions: Procedure: Type of omentectomy
- Control group/D2 radical gastrectomy with total omentectom (No Intervention): Control group with total omentectomy

INTERVENTIONS:
Procedure: Type of omentectomy — Experimental group D2 radical gastrectomy with partial omentectomy. Partial omentectomy with preservation of the greater omentum at >3 cm from the gastroepiploic arcade.Control group with total omentectomy.
  Arms: Experimental group/D2 radical gastrectomy with partial omentectomy

SUMMARY:
This is a phase III, multicenter, prospective, randomized, controlled clinical trial to evaluate the impact of omentectomy for advanced gastric cancer on patient survival.

DETAILED DESCRIPTION:
In order to evaluate the impact of omentectomy for advanced gastric cancer on patient survival, we designed this trial. Patients who received curative gastrectomy were divided into two groups based on whether they underwent omentectomy. The purpose of this study is to prove the non-inferiority of omentum preservation compared with omentectomy in patients with T3-T4a gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Had been treated with Radical resection (D2, R0) of gastric cancer (Lymph node≥16);
2. Physical condition and organ function allows to tolerable abdominal surgery;
3. Willing and able to comply with the program during the study period;
4. Written informed consent provided;
5. ≥ 18 and ≤ 70 years of age; preoperative gastric cancer patients with pathologically confirmed;
6. With more than a 6-month life expectancy;
7. No other serious concomitant diseases; Sufficient organ functions;
8. No previous history of chemotherapy or radiotherapy;
9. All patients accept 8 cycles XELOX chemotherapy regimen;
10. Clinical stage: T3-4aN0-+M0; 11 . Macroscopic types :Borrmann I-III;

12. Not greater curvature tumor; with distal or total gastrectomy； 13. No previous surgery for any abdominal disease, except an appendectomy for appendicitis, a laparoscopic cholecystectomy for gallbladder stones; No previous history of peritonitis, pancreatitis; 14. Karnofsky performance status (KPS)>60; Eastern Cooperative Oncology Group Performance Status (ECOG): 0-1.

Exclusion Criteria:

Pregnancy or breast feeding; 2. Patients with Serious liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrolled diabetes, hypertension and other chronic systemic diseases, heart disease with Clinical symptoms, such as congestive heart failure, coronary heart disease symptoms, drug is difficult to control arrhythmia, hypertension, or six months had a myocardial infarction attack, or cardiac insufficiency; 3. Organ transplantation patients need immunosuppressive therapy; 4. Severe recurrent infections were not controlled or with other serious concomitant diseases; 5. Patients got other primary malignant tumors (except curable skin basal cell carcinoma and cervical cancer in situ) except gastric cancer within 5 years; 6. Psychiatric disease which require treatment; 7. Have the history of organ transplantation; 8. Within 6 months before study starts and in the process of this study, patients participate in other clinical researches. 9. Advanced gastric cancer with omentum invasion 10. Patients can't treated with XELOX after surgery; 11 . Macroscopic types : Borrmann IV; 12. Tumor invasion of adjacent organ (T4b) or with distant metastasis#M1 #; 13. Tumor invasion the greater curvature invasion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival(DFS) | 3 years
  Disease Free Survivalof the Participants

SECONDARY OUTCOMES:
Overall Survival(OS) | 5 years
  Overall Survival of the Participants

OTHER OUTCOMES:
The volume of intraoperative blood loss | 1 week
  The volume of intraoperative blood loss (IBL) was defined as the total from suction and the weight of gauze sponges at the conclusion of the operation. The Blood loss volume is recorded in milliliters.
Postoperative morbidity | 1 month
  Postoperative morbidity was defined as the incidence rate of the postoperative complication. The postoperative morbidity were examined within 30 days after surgery. Postoperative morbidity was graded with use of the modified Clavien-Dindo classification of surgical complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastrointestinal Medical Oncology, Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No